CLINICAL TRIAL: NCT04615572
Title: Screening to Improve Survival in AL Amyloidosis
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 00000858; 1R21AG070502-01 (NIH)
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2023-11

CONDITIONS: Smoldering Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance
Keywords: SMM; MGUS; AL Amyloidosis
MeSH Terms: conditions — Smoldering Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cDNA derived from bone marrow CD138-selected plasma cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to see whether certain genes may be linked with the development of AL amyloidosis in subjects 60 years of age or older with the blood disorders SMM and MGUS. A limited repertoire of immunoglobulin (Ig) variable region genes have been associated with AL amyloidosis. The clonal plasma cells of subjects with SMM and MGUS may express one of these Ig variable region genes indicating a risk of progression to AL amyloidosis and potentially enabling early diagnosis. We hope this study will help us begin to understand whether Ig variable region gene identification can be a useful tool for assessing a subject's risk of progression to AL amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients 60 years of age and older
* Diagnosed with λ LC MGUS or λ LC SMM
* dFLC greater than 23 mg/L and κ::λ free LC ratio below normal
* If the patient has an eGFR less than 50 mL/min/1.73m2, the κ::λ free LC ratio is inconsequential. The patient only needs to meet the age, dFLC, and λ LC MGUS or λ LC SMM diagnosis criteria in this case

Exclusion Criteria:

* Patients with κ LC MGUS or κ LC SMM
* Amyloid in the bone marrow or in other biopsies will not be included
* Patients younger than 60 years of age are not eligible

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Smoldering Multiple Myeloma or Monoclonal Gammopathy of Undetermined Significance patients.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
To determine risk of AL in patients with λ SMM or λ MGUS | 2 years
  By creating a multicenter network (N =6) we will have study centers in Massachusetts (1), California (2), New York (1), North Carolina (1) and Florida (1), enabling us to evaluate 50 patients 60 or older with λ SMM or λ MGUS and to determine based on gene identification whether their clonal λ IGVL genes are AL-related. This approach will identify undiagnosed patients early in the course of AL and patients at risk for AL.
To develop a B-cell Gene Rearrangement (BCGR) test for λ IGVL germline gene identification | 2 years
  Testing for markers such as λ IGVL germline genes is highly complex as defined by the Clinical Laboratory Improvement Act (CLIA) (42 USC 263a). We will continue identifying clonal λ IGVL genes with RT-PCR using cDNA derived from bone marrow CD138-selected plasma cells in our research lab, and have partnered with a CLIA-certified diagnostic laboratory, the Columbia University Laboratory of Personalized Genomic Medicine, in order to develop and validate a next generation sequencing (NGS) approach as a CLIA compliant B-cell Gene Rearrangement Test (BCGR, CPT: 81261).
To determine if marrow mononuclear cells are adequate for λ IGVL germline gene identification | 2 years
  The multicenter trial will employ bone marrow aspirate mononuclear cells in two ways. First, a portion of each patient's marrow mononuclear cells will be used directly for cDNA for NGS and a portion used to select CD138+ plasma cells for cDNA for RT-PCR and NGS. The use of cDNA derived from bone marrow aspirate mononuclear cells for NGS would save the step of selection and be more convenient if it is equally informative. Criteria identifying specimens that likely do or do not require CD138-selection may be identified in this process.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California, Irvine Health Chao Family Comprehensive Cancer Center, Orange, California
  - University of California, San Francisco, San Francisco, California
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bodi K, Prokaeva T, Spencer B, Eberhard M, Connors LH, Seldin DC. AL-Base: a visual platform analysis tool for the study of amyloidogenic immunoglobulin light chain sequences. Amyloid. 2009 Mar;16(1):1-8. doi: 10.1080/13506120802676781. PMID 19291508
- [Background] Bujang MA, Adnan TH. Requirements for Minimum Sample Size for Sensitivity and Specificity Analysis. J Clin Diagn Res. 2016 Oct;10(10):YE01-YE06. doi: 10.7860/JCDR/2016/18129.8744. Epub 2016 Oct 1. PMID 27891446
- [Background] Comenzo RL, Wally J, Kica G, Murray J, Ericsson T, Skinner M, Zhang Y. Clonal immunoglobulin light chain variable region germline gene use in AL amyloidosis: association with dominant amyloid-related organ involvement and survival after stem cell transplantation. Br J Haematol. 1999 Sep;106(3):744-51. doi: 10.1046/j.1365-2141.1999.01591.x. PMID 10468868
- [Background] Comenzo RL, Zhang Y, Martinez C, Osman K, Herrera GA. The tropism of organ involvement in primary systemic amyloidosis: contributions of Ig V(L) germ line gene use and clonal plasma cell burden. Blood. 2001 Aug 1;98(3):714-20. doi: 10.1182/blood.v98.3.714. PMID 11468171
- [Background] Chaulagain CP, Comenzo RL. How we treat systemic light-chain amyloidosis. Clin Adv Hematol Oncol. 2015 May;13(5):315-24. PMID 26352777
- [Background] Dasari S, Theis JD, Vrana JA, Meureta OM, Quint PS, Muppa P, Zenka RM, Tschumper RC, Jelinek DF, Davila JI, Sarangi V, Kurtin PJ, Dogan A. Proteomic detection of immunoglobulin light chain variable region peptides from amyloidosis patient biopsies. J Proteome Res. 2015 Apr 3;14(4):1957-67. doi: 10.1021/acs.jproteome.5b00015. Epub 2015 Mar 20. PMID 25734799
- [Background] Dispenzieri A, Kyle RA, Katzmann JA, Therneau TM, Larson D, Benson J, Clark RJ, Melton LJ 3rd, Gertz MA, Kumar SK, Fonseca R, Jelinek DF, Rajkumar SV. Immunoglobulin free light chain ratio is an independent risk factor for progression of smoldering (asymptomatic) multiple myeloma. Blood. 2008 Jan 15;111(2):785-9. doi: 10.1182/blood-2007-08-108357. Epub 2007 Oct 17. PMID 17942755
- [Background] Dubrey SW, Cha K, Anderson J, Chamarthi B, Reisinger J, Skinner M, Falk RH. The clinical features of immunoglobulin light-chain (AL) amyloidosis with heart involvement. QJM. 1998 Feb;91(2):141-57. doi: 10.1093/qjmed/91.2.141. PMID 9578896
- [Background] Kourelis TV, Kumar SK, Go RS, Kapoor P, Kyle RA, Buadi FK, Gertz MA, Lacy MQ, Hayman SR, Leung N, Dingli D, Lust JA, Lin Y, Zeldenrust SR, Rajkumar SV, Dispenzieri A. Immunoglobulin light chain amyloidosis is diagnosed late in patients with preexisting plasma cell dyscrasias. Am J Hematol. 2014 Nov;89(11):1051-4. doi: 10.1002/ajh.23827. Epub 2014 Sep 2. PMID 25111004
- [Background] Kyle RA, Rajkumar SV. Monoclonal gammopathy of undetermined significance and smoldering multiple myeloma. Curr Hematol Malig Rep. 2010 Apr;5(2):62-9. doi: 10.1007/s11899-010-0047-9. PMID 20425398
- [Background] Kyle RA, Remstein ED, Therneau TM, Dispenzieri A, Kurtin PJ, Hodnefield JM, Larson DR, Plevak MF, Jelinek DF, Fonseca R, Melton LJ 3rd, Rajkumar SV. Clinical course and prognosis of smoldering (asymptomatic) multiple myeloma. N Engl J Med. 2007 Jun 21;356(25):2582-90. doi: 10.1056/NEJMoa070389. PMID 17582068
- [Background] Larsen JT, Kumar SK, Dispenzieri A, Kyle RA, Katzmann JA, Rajkumar SV. Serum free light chain ratio as a biomarker for high-risk smoldering multiple myeloma. Leukemia. 2013 Apr;27(4):941-6. doi: 10.1038/leu.2012.296. Epub 2012 Oct 16. PMID 23183428
- [Background] Perfetti V, Casarini S, Palladini G, Vignarelli MC, Klersy C, Diegoli M, Ascari E, Merlini G. Analysis of V(lambda)-J(lambda) expression in plasma cells from primary (AL) amyloidosis and normal bone marrow identifies 3r (lambdaIII) as a new amyloid-associated germline gene segment. Blood. 2002 Aug 1;100(3):948-53. doi: 10.1182/blood-2002-01-0114. PMID 12130507
- [Background] Perfetti V, Palladini G, Casarini S, Navazza V, Rognoni P, Obici L, Invernizzi R, Perlini S, Klersy C, Merlini G. The repertoire of lambda light chains causing predominant amyloid heart involvement and identification of a preferentially involved germline gene, IGLV1-44. Blood. 2012 Jan 5;119(1):144-50. doi: 10.1182/blood-2011-05-355784. Epub 2011 Nov 8. PMID 22067386
- [Background] Rajkumar SV, Kyle RA, Therneau TM, Melton LJ 3rd, Bradwell AR, Clark RJ, Larson DR, Plevak MF, Dispenzieri A, Katzmann JA. Serum free light chain ratio is an independent risk factor for progression in monoclonal gammopathy of undetermined significance. Blood. 2005 Aug 1;106(3):812-7. doi: 10.1182/blood-2005-03-1038. Epub 2005 Apr 26. PMID 15855274
- [Background] Tahir UA, Doros G, Kim JS, Connors LH, Seldin DC, Sam F. Predictors of Mortality in Light Chain Cardiac Amyloidosis with Heart Failure. Sci Rep. 2019 Jun 12;9(1):8552. doi: 10.1038/s41598-019-44912-x. PMID 31189919
- [Background] Zhou P, Comenzo RL, Olshen AB, Bonvini E, Koenig S, Maslak PG, Fleisher M, Hoffman J, Jhanwar S, Young JW, Nimer SD, Boruchov AM. CD32B is highly expressed on clonal plasma cells from patients with systemic light-chain amyloidosis and provides a target for monoclonal antibody-based therapy. Blood. 2008 Apr 1;111(7):3403-6. doi: 10.1182/blood-2007-11-125526. Epub 2008 Jan 23. PMID 18216299
- [Background] Zhou P, Hoffman J, Landau H, Hassoun H, Iyer L, Comenzo RL. Clonal plasma cell pathophysiology and clinical features of disease are linked to clonal plasma cell expression of cyclin D1 in systemic light-chain amyloidosis. Clin Lymphoma Myeloma Leuk. 2012 Feb;12(1):49-58. doi: 10.1016/j.clml.2011.09.217. Epub 2011 Nov 18. PMID 22100494
- [Background] Zhou P, Ma X, Iyer L, Chaulagain C, Comenzo RL. One siRNA pool targeting the lambda constant region stops lambda light-chain production and causes terminal endoplasmic reticulum stress. Blood. 2014 May 29;123(22):3440-51. doi: 10.1182/blood-2013-10-535187. Epub 2014 Apr 10. PMID 24723680